CLINICAL TRIAL: NCT07326891
Title: Continuous Glucose Monitoring in Prediabetics on a Mediterranean Diet With Sequentially Added Cycling and Rowing Training: Study Protocol for a Prospective Non-Randomized Study
Brief Title: Effects of a Mediterranean Diet With Cycling and Rowing Exercise on Blood Sugar in Women With Prediabetes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Begüm Yücesoy Güneysu (Other)
Collaborators: Marmara University (Other); Marmara University Pendik Training and Research Hospital (Other); Goztepe Prof Dr Suleyman Yalcın City Hospital (Other)
Responsible Party: Sponsor-Investigator, Begüm Yücesoy Güneysu, PhD(c), Dietitian, Principal Investigator, Marmara University
Organization: Marmara University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09.2022.946
Record Dates: First submitted 2025-12-22; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Prediabetes
Keywords: Prediabetes; Continuous Glucose Monitoring; Mediterranean Diet; Glycaemic Variability; Aerobic Exercise
MeSH Terms: conditions — Prediabetic State | interventions — Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: This is a non-randomized, three-arm, parallel-group study. Participants are allocated to one of three groups based on their glycemic status and medical eligibility for exercise: 1) Control: Mediterranean diet only (active prediabetes, exercise-ineligible); 2) Intervention Group 1: Mediterranean diet + sequential exercise (active prediabetes); 3) Intervention Group 2: Mediterranean diet + sequential exercise (prediabetes in remission). The primary scientific comparison is between the two exercise groups (Group 2 vs. Group 3) to assess the influence of baseline metabolic phenotype on intervention response.
Who Masked: Outcomes Assessor
Masking Description: Due to the behavioral nature of lifestyle interventions (supervised exercise and diet counseling), it will not be possible to blind participants or personnel administering the interventions. However, the data analyst performing the statistical analyses will be unaware of information regarding group assignment. Analysis datasets will be anonymized with neutral codes before being provided to the analyst.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): Women with medically documented prediabetes who are not eligible for the supervised exercise program for medical reasons. This arm serves as the primary comparison group and represents standard care. Participants will follow a 12-week individualized Mediterranean diet intervention emphasizing high intake of vegetables, fruits, whole grains, legumes, nuts, and olive oil; moderate consumption of fish and poultry; and low intake of red meat, processed foods, and sweets. Dietary counseling will be provided by a dietitian, and participants will complete food diaries. All participants will undergo the same scheduled assessments as the intervention arms, including blood tests, anthropometric measurements, questionnaires, and continuous glucose monitoring (CGM).
  Interventions: Other: Mediterranean Diet
- Active Prediabetes Exercise Group (Experimental): Women with active prediabetes who are medically eligible for exercise will participate in a 12-week intervention including a Mediterranean-style diet throughout the study and a supervised 8-week sequential exercise program between Weeks 3 and 10. The exercise program will consist of cycling ergometer training during Weeks 3-6 and rowing ergometer training during Weeks 7-10. Participants will complete three supervised sessions per week, each lasting approximately 51 minutes.
  Exercise intensity will be individualized using the Heart Rate Reserve (HRR) method, based on resting heart rate and maximal heart rate measured by a maximal Bruce protocol test. Each session will include a warm-up at 40% HRR, alternating intervals at 50% and 60% HRR with short recovery periods, and a cool-down at 40% HRR. Heart rate will be continuously monitored using a Polar H10 chest strap.
  Interventions: Other: Mediterranean Diet; Behavioral: Supervised Sequential Exercise
- Remission Prediabetes Exercise Group (Experimental): Participants in this arm are women with a documented diagnosis of prediabetes within the past year who are normoglycemic at screening according to American Diabetes Association (ADA) criteria and are medically eligible to participate in exercise. These participants will receive the same 12-week Mediterranean diet program and the same supervised 8-week sequential exercise intervention (cycling followed by rowing) as the active prediabetes exercise group.
  Interventions: Other: Mediterranean Diet; Behavioral: Supervised Sequential Exercise

INTERVENTIONS:
Other: Mediterranean Diet — This is a 12-week personalised dietary intervention based on the Mediterranean diet, structured around four daily meals. It emphasises a high intake of vegetables, fruits, whole grains, legumes, nuts and olive oil, as well as moderate consumption of fish and poultry, and a low intake of red meat, processed foods and sweets. Participants receive individual counselling sessions with a dietitian every two weeks and are required to keep a daily food diary to monitor adherence and provide feedback.
Behavioral: Supervised Sequential Exercise — An 8-week, supervised, sequential aerobic exercise program. Participants attend three sessions per week. The first 4 weeks consist of cycling ergometer sessions, followed by 4 weeks of rowing ergometer sessions. Exercise intensity is personalized using Heart Rate Reserve (HRR) based on directly measured maximum heart rate from a baseline cardiopulmonary exercise test. Sessions are supervised by an exercise physiologist.
  Arms: Active Prediabetes Exercise Group; Remission Prediabetes Exercise Group

SUMMARY:
The goal of this clinical trial is to learn how a Mediterranean-style diet, with and without added exercise, affects blood sugar control in women with prediabetes. Prediabetes means blood sugar levels are higher than normal but not yet type 2 diabetes. Healthy eating and regular physical activity can help prevent diabetes.

The investigators aim to answer two main questions:

1. Does adding a supervised program of cycling and rowing exercises to the diet lead to better blood sugar control than the diet alone?
2. Do women who recently returned to normal blood sugar levels respond differently to the exercise program than those who currently have high blood sugar?

Participants will be placed into one of three groups based on current blood sugar levels and medical fitness for exercise:

* Group 1 (Diet only): Will follow a Mediterranean eating plan for 12 weeks.
* Group 2 (Diet + Exercise, Current High Blood Sugar): Will follow the same diet and also do supervised exercise (cycling, then rowing) three times a week for 8 weeks.
* Group 3 (Diet + Exercise, Recent Normal Blood Sugar): Will follow the same diet and exercise program as Group 2. These women had prediabetes in the past year but now have normal blood sugar levels.

All participants will follow the study protocol for 12 weeks, which includes the following key components:

* Dietary Intervention: Adherence to a Mediterranean-style eating plan, which emphasizes high intake of vegetables, fruits, whole grains, legumes, olive oil, and fish.
* Continuous Glucose Monitoring: Wearing a continuous glucose monitoring (CGM) device-a small, minimally invasive sensor placed on the upper arm-during multiple 10-day periods. This device tracks interstitial glucose levels throughout the day and night to assess daily glucose patterns.
* Blood Sampling and Analysis: Providing fasting blood samples for the measurement of glycemic and metabolic health markers. These include fasting plasma glucose, hemoglobin A1c (HbA1c), fasting insulin, and 2-hour oral glucose tolerance test (OGTT) results.
* Anthropometric Assessments: Undergoing standardized measurements of height, body weight, body fat percentage (via bioelectrical impedance), waist circumference, and Body Mass Index (BMI) at scheduled intervals.
* Questionnaires: Completing validated surveys to assess habitual dietary intake, sleep quality and duration, and levels of physical activity.

Investigators will compare changes in blood sugar control and other health measures from the start to the end of the 12-week study among the three groups.

DETAILED DESCRIPTION:
This study aims to investigate the effects of a Mediterranean-style diet combined with cycling and rowing exercises on blood sugar control and daily blood sugar fluctuations in women with prediabetes.

Prediabetes is a condition in which blood sugar levels are higher than normal but not high enough to be diagnosed as type 2 diabetes. Importantly, prediabetes can often be reversed with appropriate lifestyle changes. Healthy eating habits and regular physical activity are the most effective ways to prevent the progression from prediabetes to diabetes. However, commonly used blood sugar tests, such as fasting glucose and hemoglobin A1c (HbA1c), do not always reflect daily ups and downs in blood sugar levels.

For this reason, this study will use continuous glucose monitoring (CGM) in addition to standard blood tests. CGM is a small sensor placed on the upper arm that measures blood sugar levels continuously throughout the day and night. This method shows how long blood sugar stays within a healthy range and how much it fluctuates during daily life. These detailed measurements allow a more accurate evaluation of how diet and exercise affect blood sugar control.

One important feature of this study is that it examines not only the effect of diet but also the effects of two different types of exercise. Participants will first perform cycling exercises, which mainly involve the lower body, and then rowing exercises, which engage both the upper and lower body. This approach allows a comparison of how different exercise types influence blood sugar regulation. In addition, evaluation will be based on metabolic background.Women whose blood sugar levels have recently returned to normal will be compared with women who still have prediabetes to determine whether responses differ to the same lifestyle program.

The study will last 12 weeks and will include three groups based on blood sugar status and medical suitability for exercise. The diet-only group will consist of women with prediabetes who are not able to participate in structured exercise for medical reasons and will follow a Mediterranean diet for 12 weeks. The diet plus exercise group will include women with ongoing prediabetes who are medically able to exercise; these participants will follow the Mediterranean diet and perform supervised exercise three times per week for 8 weeks. The third group will consist of women who were diagnosed with prediabetes within the last year but whose blood sugar levels are normal at the start of the study. This group will follow the same diet and exercise program as the second group.

The Mediterranean diet used in this study emphasizes vegetables, fruits, whole grains, legumes, olive oil, and fish, while limiting processed foods and red meat. All participants will receive individual nutrition counseling from a dietitian, and dietary adherence will be monitored regularly.

Exercise programs will be personalized for each participant. Exercise intensity will be determined using a standard exercise test performed at the beginning of the study to measure maximum heart rate. During all exercise sessions, heart rate will be continuously monitored using a chest strap to ensure safe and effective training. All exercise sessions will be conducted under professional supervision at the Faculty of Sport Sciences at Marmara University.

Throughout the study, participants' health status will be evaluated using multiple methods. The main goal is to determine how many participants achieve normal blood sugar levels by the end of the 12-week period. Blood tests will include fasting glucose, an oral glucose tolerance test (OGTT), and HbA1c. In addition, participants will wear a Dexcom G7 continuous glucose monitor during four separate 10-day periods while continuing usual daily activities.

Body weight, waist circumference, and body fat percentage will be measured at regular intervals. Sleep quality and adherence to the Mediterranean diet will be assessed using validated questionnaires.

The collected data will be analyzed to compare changes in blood sugar patterns between the different groups. Because grouping is based on existing health status rather than random assignment, the results will focus on identifying meaningful trends and individual responses rather than establishing strict cause-and-effect relationships.

At the end of this study, it is expected that clearer information will be obtained on how a Mediterranean diet combined with different types of exercise affects blood sugar control in women with prediabetes. The findings may help improve personalized lifestyle strategies for preventing diabetes and maintaining healthy blood sugar levels.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of prediabetes (within the last 1 year)

  * Impaired Fasting Glucose (IFG) 100-125 mg/dl
  * OGTT result 2-hour postprandial Impaired Glucose Tolerance (IGT) 140-199 mg/dl
  * HbA1c 5.7-6.4%
* Being between 22-55 years of age
* Being female
* Body Mass Index 18-34.9 kg/m2
* Meeting the criteria in the American College of Sports Medicine (ACSM) and American Heart Association (AHA) cardiovascular disease risk assessment scoring system
* Not engaging in regular planned exercise or physical activity (sedentary)

Exclusion Criteria:

* Diabetes
* Being pregnant
* No self-reported low iron concentrations or anaemia
* Use of medication, insulin, or weight loss injections known to affect lipid and glucose metabolism
* Presence of cardiovascular disease
* Current smoking or excessive alcohol consumption
* Presence of abnormal electrocardiogram (ECG)
* Presence of autonomic neuropathy
* Presence of uncontrolled hypertension (systolic blood pressure >135 mmHg, diastolic blood pressure >85 mmHg)
* Joint-muscle-bone injury limiting exercise

Ages: 22 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Fasting Plasma Glucose (FPG) | Baseline (week 0) and the end of the 12 weeks program (week 13)
  Change in Fasting Plasma Glucose levels, measured in mg/dL from venous blood.
Change in 2-hour Oral Glucose Tolerance Test (OGTT) Glucose | Baseline (week 0) and the end of the 12 weeks program (week 13)
  Change in plasma glucose levels measured 2 hours after a standardized glucose load, measured in mg/dL from venous blood.
Change in Hemoglobin A1c (HbA1c) | Baseline (week 0) and the end of the 12 weeks program (week 13)
  Change in the percentage (%) of glycated hemoglobin (HbA1c) measured from venous blood.
Change in Fasting Insulin | Baseline (week 0) and the end of the 12 weeks program (week 13)
  Change in fasting serum insulin levels, measured in microinternational units per milliliter (µIU/mL) from venous blood. This measurement serves as an indicator of basal insulin secretion and insulin resistance.

SECONDARY OUTCOMES:
Change in Body Weight | Baseline (Week 0), Weeks 2, 4, 6, 8, 10, and 12.
  Change in body weight measured in kilograms (kg).
Change in Body Mass Index (BMI) | Baseline (Week 0), Weeks 2, 4, 6, 8, 10, and 12.
  Weight and height measurements will be combined to report Body Mass Index in kilograms per square meter (kg/m²), calculated as weight (kg) / [height (m)]².
Change in Body Fat Percentage | Baseline (Week 0), Weeks 2, 4, 6, 8, 10, and 12.
  Change in total body fat measured as a percentage (%).
Change in Waist-to-Hip Ratio | Baseline (Week 0), Weeks 2, 4, 6, 8, 10, and 12.
  Waist and hip circumference measurements (in centimeters) will be combined to calculate and report the Waist-to-Hip Ratio. The ratio is calculated as Waist Circumference (cm) / Hip Circumference (cm) and is a unitless value. Changes in this ratio will be assessed.
Change in Glycemic Variability (CV) | Exercise groups: Baseline (week 2) , Week 6, Week 10 and Week 13. Control group: Baseline (week 2) and Week 13.
  Change in the coefficient of variation (CV, %) of glucose, a measure of daily glucose swings, measured by CGM.
Change in Continuous Glucose Monitoring (CGM)-Derived Time in Range (TIR) | First 10 days of the intervention, Last 10 days of the cycling phase (Weeks 5-6), Last 10 days of the rowing phase (Weeks 9-10), Final 10 days of the intervention.
  Change in the percentage of time spent within the target glucose range of 70-140 mg/dL, assessed using continuous glucose monitoring (CGM).
Change in Continuous Glucose Monitoring (CGM)-Derived Time Above Range (TAR) | First 10 days of the intervention, Last 10 days of the cycling phase (Weeks 5-6), Last 10 days of the rowing phase (Weeks 9-10), Final 10 days of the intervention.
  Change in the percentage of time spent with glucose levels above 140 mg/dL, assessed using continuous glucose monitoring (CGM).
Change in Continuous Glucose Monitoring (CGM)-Derived Time Below Range (TBR) | First 10 days of the intervention, Last 10 days of the cycling phase (Weeks 5-6), Last 10 days of the rowing phase (Weeks 9-10), Final 10 days of the intervention.
  Change in the percentage of time spent with glucose levels below 70 mg/dL, assessed using continuous glucose monitoring (CGM).
Change in Mean Glucose | First 10 days of the intervention, Last 10 days of the cycling phase (Weeks 5-6), Last 10 days of the rowing phase (Weeks 9-10), Final 10 days of the intervention.
  Change in the average glucose concentration, measured in mg/dL, assessed using continuous glucose monitoring (CGM).
Change in Glucose Standard Deviation (SD) | First 10 days of the intervention, Last 10 days of the cycling phase (Weeks 5-6), Last 10 days of the rowing phase (Weeks 9-10), Final 10 days of the intervention.
  Description: Change in the standard deviation (SD) of glucose values, measured in mg/dL. The SD is calculated as the root mean square of the deviation of all CGM-measured glucose values from their mean over a specified period, representing the absolute variability of glucose concentrations.
Change in Coefficient of Variation (CV) | First 10 days of the intervention, Last 10 days of the cycling phase (Weeks 5-6), Last 10 days of the rowing phase (Weeks 9-10), Final 10 days of the intervention.
  Change in the coefficient of variation (CV) of glucose values, expressed as a percentage (%). The CV is calculated for a specified period as: (Standard Deviation of Glucose / Mean Glucose) × 100. This metric represents the relative glycemic variability, normalized to the individual's mean glucose level, as assessed by continuous glucose monitoring (CGM).
Change in Glucose Management Indicator (GMI) | First 10 days of the intervention, Last 10 days of the cycling phase (Weeks 5-6), Last 10 days of the rowing phase (Weeks 9-10), Final 10 days of the intervention.
  Change in the estimated average glucose level expressed as a percentage (%), calculated from CGM data, which correlates with the laboratory hemoglobin A1c (HbA1c) measure.
Change in Area Under the Curve (AUC) for Glucose | First 10 days of the intervention, Last 10 days of the cycling phase (Weeks 5-6), Last 10 days of the rowing phase (Weeks 9-10), Final 10 days of the intervention.
  Change in the total area under the glucose curve, measured in mg·h/dL, assessed over specified periods using continuous glucose monitoring (CGM).
Change in Mediterranean Diet Adherence (MEDAS Score) | Baseline (week 0) and the end of the 12 weeks program (week 13)
  Change in adherence to the diet, measured by the 14-item Mediterranean Diet Adherence Scale (MEDAS). Total scores range from 0 to 14, with higher scores indicating better adherence.
Change in Sleep Quality (PSQI) | Baseline (week 0) and the end of the 12 weeks program (week 13)
  Change in sleep quality measured by the Pittsburgh Sleep Quality Index. Scores range 0-21 (lower = better).

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Birol Çotuk, Prof., Study Director — Turkish-German University
Locations (1):
- Marmara University, Beykoz, Istanbul, Turkey (Türkiye)